CLINICAL TRIAL: NCT05286736
Title: Plasticity of Motor Systems in Early Stage Parkinson's Disease
Brief Title: Neuroplasticity in Parkinson's Disease
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: NEUR-2019-28388
Record Dates: First submitted 2022-02-17; First posted 2022-03-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Parkinson; Parkinson Disease
Keywords: Parkinson's
MeSH Terms: conditions — Parkinson Disease | interventions — Neuroimaging

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- Early (untreated) Parkinson's Disease: Diagnosis of idiopathic PD, as determined by a movement disorders neurologist in accordance with the PD Society Brain Bank diagnostic criteria.
  Interventions: Diagnostic Test: Neuroimaging; Diagnostic Test: Quantitative assessments
- Healthy Controls: Age- and sex-matched healthy controls.
  Interventions: Diagnostic Test: Neuroimaging; Diagnostic Test: Quantitative assessments

INTERVENTIONS:
Diagnostic Test: Neuroimaging — This project will use neuroimaging (7T MRI: structural, diffusion and rest-state functional MRI) and non-invasive brain stimulation (TMS: PAS. SAI) techniques to quantify structural and functional changes in brain function.
Diagnostic Test: Quantitative assessments — Quantitative assessments of motor function (gait, gait initiation, reactive balance, bradykinesia, repetitive alternating movements, rigidity, stop-signal reaction time), and neuropsychological function

SUMMARY:
The purpose of this project is to increase our understanding of the early state and temporal evolution of neuroplastic changes in the cortex and subthalamic nucleus (STN) of people with PD, and the relationship of these changes to the emergence and expression of PD motor and non-motor signs. Neurophysiological biomarkers derived from this work may be important for the early detection and prediction of progression of disease. They can also provide the means to assess the efficacy of interventions designed to prevent or slow disease progression.

DETAILED DESCRIPTION:
This project will use neuroimaging (7T MRI: structural, diffusion and rest-state functional MRI), from Dr. Noam Harel's protocol IRB# STUDY00008096, and non-invasive brain stimulation (TMS: PAS. SAI) techniques to quantify structural and functional changes in brain function. The TMS experiment will use a Magstim Bistimn 2002 transcranial magnetic stimulation (TMS) unit and standard figure-of-eight coil (70 mm diameter) to deliver stimulation on the surface of the scalp. Stimulation will be delivered using either a single pulse or with a paired-pulse protocol (two stimuli, through the same TMS coil at inter-stimulus intervals of 50 or 80 ms). All surface EMG signals will be pre-amplified within the sensor and sent wirelessly via blue-tooth connection to a Delsys data collection system. Quantitative assessments of motor function (gait, gait initiation, reactive balance, bradykinesia, repetitive alternating movements, rigidity, stop-signal reaction time), and neuropsychological function will used to assess behavioral status at baseline and 30-36 months later.

ELIGIBILITY:
Inclusion Criteria:

Participants with PD

* Diagnosis of idiopathic PD, as determined by a movement disorders neurologist in accordance with the PD Society Brain Bank diagnostic criteria
* Not receiving levodopa or dopamine agonist to treat PD (at baseline)
* Able to ambulate independently without the use of an assistive device (e.g. cane) for 50 meters Healthy Controls
* Age- (+/- 3 years) and sex-matched to participants with PD
* Able to ambulate independently without the use of an assistive device (e.g. cane) for 50 meters

Exclusion Criteria:

* Dementia diagnosis and/or a University of California Brief Assessment of Capacity to Consent (UBACC) score and MacCAT-CR score indicating impaired capacity to consent
* History of musculoskeletal disorders that significant affect movement of lower or upper limbs as determined at the time of enrollment
* History of bipolar disorder, post-traumatic stress disorder or major depressive disorder
* Other significant neurological disorders that may affect participation or performance in the study
* Implanted DBS or other neurosurgeries to treat PD
* Pregnancy

Additional exclusion criteria for TMS experiments (note that individuals who are excluded from the TMS experiment still have the opportunity to participate in the other data collection sessions):

* History of seizures, epilepsy, stroke, multiple sclerosis, or traumatic brain injury
* Recent history of frequent syncope (fainting) episodes in response to blood, emotional stress, or sensory triggers.
* Intracranial metallic or magnetic devices (e.g. cochlear implant, deep brain stimulator)
* Pacemaker or any implanted device
* History of surgery on blood vessels, brain, or heart
* Unexplained, recurring headaches or concussion within the last six months
* Severe hearing impairment

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Parkinson's Disease (early diagnosis, currently untreated) and age- and sex-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2026-07-09 (Estimated); Study Completion 2028-11-09 (Estimated)

PRIMARY OUTCOMES:
Change in volume of Subthalamic Nucleus | Baseline, 30-36 months
  The volume of the subthalamic nucleus is assessed using MRI and reported in millimeters cubed (mm^3).
Change in fractional Anisotropy of Subthalamic Nucleus | Baseline, 30-36 months
  Fractional anisotropy, measured using MRI, is a unit-less value between zero and one that describes the degree of anisotropy of water diffusion in a specified brain area. Higher values indicate a greater degree of anisotropy, while a score of zero indicates isotropic diffusion.
Change in cortico-STN Connectivity | Baseline, 30-36 months
  Cortico-Subthalamic nucleus connectivity is measured using MRI and reported as a z score (unitless).
Change in paired Associative Stimulation-Motor Evoked Potential (PAS-MEP) | Baseline, 30-36 months
  Motor evoked potential is measured as the amplitude of change in target muscle electrical activity following transcranial magnetic stimulation (TMS) and reported in units of millivolts (mV).
Change in Mattis Dementia Rating Scale 2 (DRS-2) | Baseline, 30-36 months
  The DRS-2 consists of 24 items, rated on a scale from 0 to 6. Item scores are combined into five subscales: attention (8 items), initiation/perseveration (11 items), construction (6 items), conceptualization ( 6 items), and memory (5 items). These five subscale scores are summed to calculate a total score ranging from from 0 to 144 points, with lower scores indicating worse performance due to dementia.
Change in Rey Complex Figure and Matrix Reasoning of the Wechsler Adult Intelligence Scale - IV | Baseline, 30-36 months
Change in Stroop Color Word Test | Baseline, 30-36 months
Change in Wisconsin Card Sorting Test | Baseline, 30-36 months
Change in Delis-Kaplan Executive Function System (D-KEFS) Verbal Fluency Subtest | Baseline, 30-36 months
Change in Brief Visuospatial Memory Test - Revised (BVMT-R) | Baseline, 30-36 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States